CLINICAL TRIAL: NCT02832921
Title: Cognitive-motor Intervention Using Virtual Reality for Middle-aged Individuals at High Dementia Risk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SHEBA-16-2988-MSB-CTIL
Record Dates: First submitted 2016-06-26; First posted 2016-07-14 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Alzheimer's Disease (AD)
Keywords: Alzheimer's disease; virtual reality; cognitive training
MeSH Terms: conditions — Alzheimer Disease | interventions — Exercise Test

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- VR cognitive tasks + treadmill (Experimental): This is the primary group of interest, in which the investigators hypothesize the greatest cognitive gains since motor activity will augment cognitive activity.
  Interventions: Behavioral: cognitive training by virtual reality; Device: treadmill
- VR cognitive tasks - treadmill (Active Comparator): This group will be an active control, receiving the VR cognitive training without treadmill walking, to examine whether the motor component augments the effect of the VR in the experimental group.
  Interventions: Behavioral: cognitive training by virtual reality
- scientific TV documentary + treadmill (Sham Comparator): This group will watch a scientific TV documentary while walking on the treadmill. This control group will permit examination of whether the VR cognitive training, which requires an especially active cognitive effort while walking on the treadmill, is more advantageous than passively watching a scientific TV documentary while performing the same motor task as the experimental group.
  Interventions: Behavioral: watching a scientific TV documentary; Device: treadmill
- Passive control (No Intervention): This group of participants will not receive any intervention but will be assessed with the same battery of assessments as the other three groups, permitting comparisons of the cognitive and neurobiological outcomes of the intervention groups to that of the natural course of decline/deterioration of these at-risk individuals.

INTERVENTIONS:
Behavioral: cognitive training by virtual reality
  Arms: VR cognitive tasks + treadmill; VR cognitive tasks - treadmill
Behavioral: watching a scientific TV documentary
  Arms: scientific TV documentary + treadmill
Device: treadmill — VR cognitive training will be augmented by walking on a treadmill, since it is well established that dual tasking-i.e. performing the VR-based cognitive effort together with a motor task, even as simple as walking on a treadmill-places greater demand on cognitive resources than a "single task".
  Arms: VR cognitive tasks + treadmill; scientific TV documentary + treadmill

SUMMARY:
The primary objective of this program is to apply a virtual reality (VR) cognitive-motor intervention (compared to active and passive control groups) to delay or slow cognitive decline of middle-aged adults who have a family history of Alzheimer's disease (AD) and thus are at particularly high risk of developing the disease.

ELIGIBILITY:
Inclusion Criteria:

* The participants of the study must have at least one parent with Alzheimer's disease.
* Fluency in Hebrew, in order to understand the instructions of the cognitive tests.
* Availability of an informant for the participant.

Exclusion Criteria:

* Severe neurological or psychological conditions that may affect cognitive performance.
* Substantial orthopedic limitations which prevent the use of treadmill.
* Unstable medical condition such as an active cancer.
* Incapability of adherence to the training program.
* The participant is undergoing a treatment that may interfere with the study program.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-07 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
change in overall cognition- measured by averaging z-scores from 14 paper and pencil neuropsychological tests covering episodic memory and executive functions cognitive domains. | baseline, immediately after 12-week training, and 3 months post-training (or corresponding time points in passive control group)
  summary of the z-scores of all 14 paper and pencil cognitive tests
change in cerebral blood flow from arterial spin labeling (ASL) | baseline, immediately after 12-week training, and 3 months post-training (or corresponding time points in passive control group)
  acquired by structural MRI using background-suppressed pseudo-continuous ASL (pcASL) featuring a 3D fast spin echo spiral sequence

SECONDARY OUTCOMES:
specific cognitive domains- average of z-scores of paper and pencil memory tests and of executive functions tests | baseline, immediately after 12-week training, and 3 months post-training (or corresponding time points in passive control group)
  summary of z-scores of executive functions tests and of episodic memory tests
blood oxygenation level dependent (BOLD) functional MRI (fMRI) signal in the fronto-parietal network associated with working memory | baseline, immediately after 12-week training, and 3 months post-training (or corresponding time points in passive control group)
  T2*-weighted fMRI during an n-back working memory task; contrasts: 1-back minus 0-back; 2-back minus 0-back; 2-back minus 1-back
brain resting state functional connectivity by resting state network fMRI BOLD signal correlations | baseline, immediately after 12-week training, and 3 months post-training (or corresponding time points in passive control group)
  T2*-weighted fMRI while relaxing with eyes closed; functional connectivity between seed regions of resting state networks (e.g., default mode, attentional, salience) and other regions by correlation of BOLD signal in seed regions with that in other regions
hippocampal volume | baseline, immediately after 12-week training, and 3 months post-training (or corresponding time points in passive control group)
  3D T1-weighted MRI imaging
frontal inferior cortex volume | baseline, immediately after 12-week training, and 3 months post-training (or corresponding time points in passive control group)
  3D T1-weighted MRI imaging
white matter hyperintensity (WMH) burden | baseline, immediately after 12-week training, and 3 months post-training (or corresponding time points in passive control group)
  3D T2-FLAIR MRI imaging
diffusion-tensor imaging (DTI) measures | baseline, immediately after 12-week training, and 3 months post-training (or corresponding time points in passive control group)
  diffusion-weighted MRI imaging (DWI) to map white matter tractography

CONTACTS AND LOCATIONS:
Overall Officials: Michal Schnaider Beeri, PhD, Principal Investigator — Sheba Medical Center/Icahn School of Medicine at Mount Sinai
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garthe A, Roeder I, Kempermann G. Mice in an enriched environment learn more flexibly because of adult hippocampal neurogenesis. Hippocampus. 2016 Feb;26(2):261-71. doi: 10.1002/hipo.22520. Epub 2015 Sep 15. PMID 26311488
- [Background] Lazarov O, Robinson J, Tang YP, Hairston IS, Korade-Mirnics Z, Lee VM, Hersh LB, Sapolsky RM, Mirnics K, Sisodia SS. Environmental enrichment reduces Abeta levels and amyloid deposition in transgenic mice. Cell. 2005 Mar 11;120(5):701-13. doi: 10.1016/j.cell.2005.01.015. PMID 15766532
- [Background] Gould E, Reeves AJ, Fallah M, Tanapat P, Gross CG, Fuchs E. Hippocampal neurogenesis in adult Old World primates. Proc Natl Acad Sci U S A. 1999 Apr 27;96(9):5263-7. doi: 10.1073/pnas.96.9.5263. PMID 10220454
- [Background] Gould E, Reeves AJ, Graziano MS, Gross CG. Neurogenesis in the neocortex of adult primates. Science. 1999 Oct 15;286(5439):548-52. doi: 10.1126/science.286.5439.548. PMID 10521353
- [Background] Stern Y. Cognitive reserve in ageing and Alzheimer's disease. Lancet Neurol. 2012 Nov;11(11):1006-12. doi: 10.1016/S1474-4422(12)70191-6. PMID 23079557
- [Background] Esiri MM, Chance SA. Cognitive reserve, cortical plasticity and resistance to Alzheimer's disease. Alzheimers Res Ther. 2012 Mar 1;4(2):7. doi: 10.1186/alzrt105. PMID 22380508
- [Background] Gaitan A, Garolera M, Cerulla N, Chico G, Rodriguez-Querol M, Canela-Soler J. Efficacy of an adjunctive computer-based cognitive training program in amnestic mild cognitive impairment and Alzheimer's disease: a single-blind, randomized clinical trial. Int J Geriatr Psychiatry. 2013 Jan;28(1):91-9. doi: 10.1002/gps.3794. Epub 2012 Apr 3. PMID 22473855
- [Background] Gates NJ, Valenzuela M, Sachdev PS, Singh NA, Baune BT, Brodaty H, Suo C, Jain N, Wilson GC, Wang Y, Baker MK, Williamson D, Foroughi N, Fiatarone Singh MA. Study of Mental Activity and Regular Training (SMART) in at risk individuals: a randomised double blind, sham controlled, longitudinal trial. BMC Geriatr. 2011 Apr 21;11:19. doi: 10.1186/1471-2318-11-19. PMID 21510896
- [Background] Rebok GW, Ball K, Guey LT, Jones RN, Kim HY, King JW, Marsiske M, Morris JN, Tennstedt SL, Unverzagt FW, Willis SL; ACTIVE Study Group. Ten-year effects of the advanced cognitive training for independent and vital elderly cognitive training trial on cognition and everyday functioning in older adults. J Am Geriatr Soc. 2014 Jan;62(1):16-24. doi: 10.1111/jgs.12607. Epub 2014 Jan 13. PMID 24417410
- [Background] Hausdorff JM, Schweiger A, Herman T, Yogev-Seligmann G, Giladi N. Dual-task decrements in gait: contributing factors among healthy older adults. J Gerontol A Biol Sci Med Sci. 2008 Dec;63(12):1335-43. doi: 10.1093/gerona/63.12.1335. PMID 19126846
- [Background] Optale G, Urgesi C, Busato V, Marin S, Piron L, Priftis K, Gamberini L, Capodieci S, Bordin A. Controlling memory impairment in elderly adults using virtual reality memory training: a randomized controlled pilot study. Neurorehabil Neural Repair. 2010 May;24(4):348-57. doi: 10.1177/1545968309353328. Epub 2009 Nov 24. PMID 19934445
- [Background] Man DW, Chung JC, Lee GY. Evaluation of a virtual reality-based memory training programme for Hong Kong Chinese older adults with questionable dementia: a pilot study. Int J Geriatr Psychiatry. 2012 May;27(5):513-20. doi: 10.1002/gps.2746. Epub 2011 Jun 17. PMID 21681818
- [Background] Tarraga L, Boada M, Modinos G, Espinosa A, Diego S, Morera A, Guitart M, Balcells J, Lopez OL, Becker JT. A randomised pilot study to assess the efficacy of an interactive, multimedia tool of cognitive stimulation in Alzheimer's disease. J Neurol Neurosurg Psychiatry. 2006 Oct;77(10):1116-21. doi: 10.1136/jnnp.2005.086074. Epub 2006 Jul 4. PMID 16820420
- [Background] Birdsill AC, Carlsson CM, Willette AA, Okonkwo OC, Johnson SC, Xu G, Oh JM, Gallagher CL, Koscik RL, Jonaitis EM, Hermann BP, LaRue A, Rowley HA, Asthana S, Sager MA, Bendlin BB. Low cerebral blood flow is associated with lower memory function in metabolic syndrome. Obesity (Silver Spring). 2013 Jul;21(7):1313-20. doi: 10.1002/oby.20170. Epub 2013 May 19. PMID 23687103
- [Background] Gommer ED, Martens EG, Aalten P, Shijaku E, Verhey FR, Mess WH, Ramakers IH, Reulen JP. Dynamic cerebral autoregulation in subjects with Alzheimer's disease, mild cognitive impairment, and controls: evidence for increased peripheral vascular resistance with possible predictive value. J Alzheimers Dis. 2012;30(4):805-13. doi: 10.3233/JAD-2012-111628. PMID 22460326
- [Background] Beeri MS, Ravona-Springer R, Moshier E, Schmeidler J, Godbold J, Karpati T, Leroith D, Koifman K, Kravitz E, Price R, Hoffman H, Silverman JM, Heymann A. The Israel Diabetes and Cognitive Decline (IDCD) study: Design and baseline characteristics. Alzheimers Dement. 2014 Nov;10(6):769-78. doi: 10.1016/j.jalz.2014.06.002. Epub 2014 Aug 20. PMID 25150735
- [Background] Villemagne VL, Burnham S, Bourgeat P, Brown B, Ellis KA, Salvado O, Szoeke C, Macaulay SL, Martins R, Maruff P, Ames D, Rowe CC, Masters CL; Australian Imaging Biomarkers and Lifestyle (AIBL) Research Group. Amyloid beta deposition, neurodegeneration, and cognitive decline in sporadic Alzheimer's disease: a prospective cohort study. Lancet Neurol. 2013 Apr;12(4):357-67. doi: 10.1016/S1474-4422(13)70044-9. Epub 2013 Mar 8. PMID 23477989
- [Background] Bauckneht M, Picco A, Nobili F, Morbelli S. Amyloid positron emission tomography and cognitive reserve. World J Radiol. 2015 Dec 28;7(12):475-83. doi: 10.4329/wjr.v7.i12.475. PMID 26753062
- [Background] Van der Mussele S, Fransen E, Struyfs H, Luyckx J, Marien P, Saerens J, Somers N, Goeman J, De Deyn PP, Engelborghs S. Depression in mild cognitive impairment is associated with progression to Alzheimer's disease: a longitudinal study. J Alzheimers Dis. 2014;42(4):1239-50. doi: 10.3233/JAD-140405. PMID 25024328